CLINICAL TRIAL: NCT00825240
Title: Formative Study of Tailored Survivor Health Promotion
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0296
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Cancer Survivorship Study; Questionnaires; Survivorship; Survivor Health; Health Promotion; Behavior Changes; Computer-assisted intervention program
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Survivorship Study: Survey of colorectal cancer patients within one year from treatment end.
  Interventions: Behavioral: One-time Questionnaire + Recorded Qualitative Interview

INTERVENTIONS:
Behavioral: One-time Questionnaire + Recorded Qualitative Interview — One-time questionnaire + recorded qualitative interview, approximately 45 minutes total.
  Other Names: surveys

SUMMARY:
The overall goal of this study is to explore colorectal cancer patients' concerns and interest about their health and behavior changes post treatment. Investigators will conduct formative research, which includes qualitative interviews, to assess the issues that cancer survivors are willing to work on as they transition out of active treatment.

The specific aims are as follows:

Aim 1: Use qualitative interview methods to describe the taxonomy of domains health promotion and illness prevention behavior changes for which colorectal cancer survivors need new information, skills training and support.

Aim 2: Explore colorectal cancer patients' perceptions of their post treatment functional status.

Aim 3: Explore the impact of cancer, treatment, and co-morbidities on colorectal cancer patients' health goals and functional status.

DETAILED DESCRIPTION:
Study Procedures:

If you agree to take part in this study, you will be asked to fill out a questionnaire about the your current health status, social support and goals.

After completing the questionnaire, you will have an interview with a research assistant. The interview will be audio recorded. You will be asked about goals you have for your health, what you are doing to reach those goals, resources you would like to receive, and challenges you faced since completing your treatment.

Your name and any of your other personal identifying information will not be linked to or collected with any of your responses. All audio tapes will be destroyed at the end of the study.

Length of Study :

The total time of participation for this study is about 45 minutes.

This is an investigational study. Up to 45 patients will be enrolled in this multicenter study. Up to 15 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with Stage IIB or III colorectal cancer.
2. Men and women within 1 year of ending primary treatment for colorectal cancer.
3. Over 18 years of age.
4. Must be able to read and write English.
5. Must be able to understand and provide written informed consent.

Exclusion Criteria:

1) Patients who have had previous treatment for cancer before treatment at M.D. Anderson, Kelsey-Seybold, and the VA Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IIB or III Colorectal cancer patients over 18 years of age ending cancer treatment or have completed cancer treatment.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Patients' Concerns + Behavior Changes Post Treatment | Qualitative data collection over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Holly Holmes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Kelsey Research Foundation, Houston, Texas
  - The Michael E. DeBakey VA Medical Center, Baylor College of Medicine, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org